CLINICAL TRIAL: NCT00011037
Title: A Multisite Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of ALVAC-HIV vCP1452 Alone and Combined With MN rgp120
Brief Title: ALVAC-HIV vCP1452 Alone and Combined With MN rgp120
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 026/HIVNET 026; 10529 (Registry Identifier: DAIDS ES Registry Number); HIVNET 026
Record Dates: First submitted 2001-02-08; First posted 2001-08-31 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: HIV Antibodies; HIV Antigens; HIV Envelope Protein gp120; AIDS Vaccines; CD4-Positive T-Lymphocytes; CD8-Positive T-Lymphocytes; Neutralization Tests; Haiti; Brazil; Cytotoxicity, Immunologic; Epitopes; Viral Proteins; Trinidad and Tobago; Peru; HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- 1 (Experimental): Participants will receive ALVAC-HIV vCP1452 at 0, 1, 3, and 6 months and MN rgp120 and Months 3 and 6
  Interventions: Biological: ALVAC(2)120(B,MN)GNP (vCP1452); Biological: MN rgp120/HIV-1
- 2 (Experimental): Participants will receive ALVAC-HIV vCP1452 at 0, 1, 3, and 6 months and MN rgp120 placebo and Months 3 and 6
  Interventions: Biological: ALVAC(2)120(B,MN)GNP (vCP1452); Biological: MN rgp120/HIV-1 placebo
- 3 (Placebo Comparator): Participants will receive ALVAC-HIV vCP1452 placebo at 0, 1, 3, and 6 months and MN rgp120 placebo and Months 3 and 6
  Interventions: Biological: ALVAC(2)120(B,MN)GNP (vCP1452) placebo; Biological: MN rgp120/HIV-1 placebo

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452) — 1 x 10^ 7 TCID50 administered intramuscularly
  Arms: 1; 2
Biological: MN rgp120/HIV-1 — 0.6 mg administered intramuscularly
  Arms: 1
Biological: ALVAC(2)120(B,MN)GNP (vCP1452) placebo — ALVAC placebo administered intramuscularly
  Arms: 3
Biological: MN rgp120/HIV-1 placebo — Alum placebo administered intramuscularly
  Arms: 2; 3

SUMMARY:
The purpose of this study is to test how the body's immune system responds to the vaccine ALVAC-HIV vCP1452 and to determine if the vaccine is safe when given alone and with MN rgp120.

HIV infection and AIDS have no cure, in spite of recent advances in anti-HIV drugs. Many worldwide populations cannot afford the antiviral treatments for infected people. HIV vaccines offer hope for disease prevention. In this trial, 2 experimental HIV vaccines called ALVAC vCP1452 and MN rgp120 will be given to volunteers in Haiti, Brazil, Peru, and Trinidad and Tobago. The study will determine how volunteers' immune systems respond to the vaccines. (This protocol has been changed by adding new international sites.)

DETAILED DESCRIPTION:
There is no cure for HIV infection or AIDS in spite of recent advances in antiviral therapy. Furthermore, drug therapy is too expensive for most affected populations. For this reason, there is a commitment to the development of safe, effective vaccines to prevent HIV infection and AIDS worldwide. This study evaluates the immunogenicity and safety of candidate HIV-1 vaccines, based on the canarypox vector termed ALVAC, alone and combined with an MN rgp120 product, at 3 [AS PER AMENDMENT 7/19/01: 5] international sites.

[AS PER AMENDMENT 7/19/01: Volunteers in Rio de Janeiro, Haiti, and Trinidad and Tobago comprise Part I; volunteers in Sao Paulo and Peru comprise Part II.] Volunteers from Haiti, Brazil, [AS PER AMENDMENT 7/19/01: Peru] and Trinidad and Tobago are enrolled into 1 of 3 arms and followed for 18 months. Arm 1 volunteers receive ALVAC-HIV vCP1452 at 0, 1, 3, and 6 months. Arm 2 volunteers receive ALVAC-HIV vCP1452 on the same schedule as Arm 1 and receive HIV-1 MN rgp120 subunit simultaneously with the 3-month and 6-month vaccine doses. Arm 3 volunteers receive a placebo. Blood and urine samples are collected for immunologic assays, virologic determinations, pregnancy testing, and safety assessments. Risk behavior and social harms are assessed every 6 months during follow-up [AS PER AMENDMENT 7/19/01: Social harms are assessed every 3 months during follow-up and risk behavior every 6 months]. At all clinic visits volunteers receive counseling on avoidance of HIV infection and pregnancy. Participants are tested for HIV-1 every 3 [AS PER AMENDMENT 7/19/01: the following text has been deleted: to 6] months. Counseling and follow-up for any needed medical care are provided.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are from Brazil (Rio de Janeiro), Haiti, Peru, or Trinidad and Tobago.
* Are 18 to 60 years old.
* Are HIV-negative.
* Have not developed a sexually transmitted disease in the last 6 months.
* Have had no more than 2 sexual partners in the last 6 months.
* Have not injected drugs or used crack cocaine in the last 6 months.
* Have not exchanged sex for money or drugs in the last 6 months.
* Have used an adequate birth control method for 1 month prior to study injections and intend to continue for the injection period (7 months).
* Are available for 18 months of follow-up.
* Have a normal history and physical examination.
* (The criteria for inclusion have been changed from the original.)

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Have had immune diseases, chronic illness, or cancer (unless cured by surgical removal), or have used medications affecting the immune system.
* Have a medical or mental condition, or job that interferes with the study requirements.
* Have a sexual partner who is HIV-infected, unless practicing abstinence or have always used condoms for the last 6 months.
* Have a sexual partner at high risk of HIV infection.
* Have received live vaccines or experimental agents within 30 days prior to planned vaccination.
* Have received blood products or immunoglobulin in the past 6 months.
* Have active tuberculosis.
* Have had a severe allergic reaction, including 1 requiring hospitalization or medical care, or a serious reaction to vaccines.
* Have received HIV-1 vaccines or placebo in a previous HIV vaccine trial.
* Are pregnant or breast-feeding.
* Are allergic to egg products, thimerosal, or neomycin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity and safety of two vaccine regimens | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wright, Study Chair
Locations (4):
- Projeto Praça Onze/Hesfa Crs, Rio de Janeiro, Brazil
- Les Centres GHESKIO CRS, Port-au-Prince, Haiti
- Barranco CRS, Lima, Peru
- CCPRI Med. Ctr. - Med. Research Foundation of Trinidad & Tobago, Port of Spain, Trinidad and Tobago